CLINICAL TRIAL: NCT00828815
Title: A Phase I, Open-label Trial to Investigate the Pharmacokinetic Effect of Multiple-dose TMC125 on Buprenorphine and Norbuprenorphine Administered in HIV-negative Subjects on Stable Buprenorphine/Naloxone Maintenance Therapy.
Brief Title: TMC125-TiDP2-C188: A Phase I, Open-label Trial to Investigate the Pharmacokinetic Effect of Multiple-dose TMC125 on Buprenorphine and Norbuprenorphine Administered in HIV-negative Patients on Stable Buprenorphine/Naloxone Maintenance Therapy.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015775
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-10

CONDITIONS: HIV; Pharmacokinetics
Keywords: HIV-negative; buprenorphine/nalaxone; norbuprenorphine; opioid-dependent; TMC125-TiDP2-C188; TMC125-C188; TMC125; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
TMC125 is from the class of drugs called non-nucleoside reverse transcriptase inhibitors (NNRTIs). NNRTIs work by blocking reverse transcriptase, a protein that HIV needs to make more copies of itself. TMC125 is used in the treatment of adults with HIV-1 infection. The purpose of this trial is to see if there is any potential interaction (change in the effectiveness of the drug) when taking multiple-dose TMC125 and buprenorphine/naloxone together. The trial will also assess the short-term safety and tolerability (how well your body handles the drug) when TMC125 and buprenorphine/naloxone are taken together.

DETAILED DESCRIPTION:
This is a Phase I, open-label (patient and trial doctor know what medication you are taking at any point in time during the trial), add-on trial in patients who are on stable sublingual (placed in the mouth under the tongue until it disolves) buprenorphine/naloxone maintenance therapy, to investigate the potential pharmacokinetic effect of multiple-dose TMC125 on buprenorphine and norbuprenorphine administered as buprenorphine/naloxone. The study population will consist of 16 HIV-negative opioid-dependent patients on stable individualized sublingual buprenorphine/naloxone maintenance therapy. Patients will first participate in a 2 weeks run-in period with supervised buprenorphine/naloxone intake. Subsequently, patients will receive TMC125 200 mg orally twice daily for 14 days added to their buprenorphine/naloxone treatment. During the treatment period from Day 1 to Day 14, the individualized buprenorphine/naloxone treatment will be continued with co-administration of TMC125. Full pharmacokinetic profiles of buprenorphine and norbuprenorphine will be determined on Days -1 and 14 up to 24 hours postdose. Full pharmacokinetic profiles of TMC125 will be determined on Day 14 up to 12 hours postdose. Pharmacodynamic assessments of symptoms of opiate withdrawal and excess will be performed. The short-term safety and tolerability will be assessed throughout the trial. Patients will firstparticipate in a 2 weeks run-in period with supervised buprenorphine/naloxone intake. Subsequently, patients will receive 2 tablets of 100 mg TMC125 twice daily for 14 days added to their buprenorphine/naloxone treatment. During the treatment period from Day 1 to Day 14, the individualized buprenorphine/naloxone treatment will be continued with co-administration of TMC125.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, extremes included. BMI is calculated as the weight (in kg) divided by the square of height (in m)
* Receiving once daily buprenorphine/naloxone maintenance therapy at a stable individualized dose formulated and administered as sublingual tablets with a maximum daily dose of 16/4 mg of buprenorphine/naloxone. Patients using buprenorphine only are also eligible if they switch to buprenorphine/naloxone minimally 2 weeks before randomization
* The patient agrees not to change the current buprenorphine/naloxone therapy from Screening until Day 14 included (switching buprenorphine to buprenorphine/naloxone between Screening and Day -14 is allowed)and to have a daily observed and documented buprenorphine/naloxone intake from Day -14 until Day 15
* General medical condition, in the investigator's opinion, does not interfere with the assessments and the completion of the trial.

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test at Screening
* Female, except if postmenopausal since more than 2 years, or posthysterectomy, or post-tubal ligation (without reversal operation)
* Evidence of current use of barbiturate, amphetamine, recreational or narcotic drug use (cocaine, inhalants, stimulants), sedative hypnotics (benzodiazepines), excessive alcohol or opioids. The drug screening involves analysis for amphetamines, barbiturates, benzodiazepines, cocaine and opioids
* Hepatitis A infection (confirmed by hepatitis A antibody IgM), or hepatitis B infection (confirmed by hepatitis B surface antigen) at study screening
* Currently active gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the effect of multiple-dose TMC125 on the steady-state pharmacokinetics of buprenorphine and its metabolite norbuprenorphine in HIV-negative patients during 2 weeks.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of TMC125, the pharmacodynamic effects of opiate excess or withdrawal and short-term safety and tolerability of the co-administration of TMC125 and buprenorphine/naloxone during 2 weeks of coadministration with TMC125.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: A Phase I, open-label study to investigate the pharmacokinetic effects of multiple-dose etravirine onbuprenorphine and norbuprenorphine administered in HIV-negative subjects on stablebuprenorphine/naloxone maintenance therapy. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1018&filename=CR015775_CSR.pdf